CLINICAL TRIAL: NCT05069246
Title: The Clinical Assessment of Nigella Sativa Oil vs Chlorohexidine as a Therapeutic Aid for Gingivitis, Effect on Gingival IL-6 and IL-18 and Antimicrobial Efficacy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ishrat Rahman (Other)
Responsible Party: Sponsor-Investigator, Ishrat Rahman, Assistant Professor, Princess Nourah Bint Abdulrahman University
Organization: Princess Nourah Bint Abdulrahman University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNU-IRB: 20-0261
Record Dates: First submitted 2021-09-18; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Nigella sativa oil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 / Nigella Sativa oil / NS (Experimental): Group 1- Nigella Sativa (NS) N. sativa oil (Al-Hussan Food Products Factory, Riyadh, Kingdom of Saudi Arabia), which was brought from the local market in Riyadh.
  Each participant was given a 3 weeks supply of oil, and a sterile plastic 15ml graduated measuring cap. They were asked to measure 5ml of oil into the cap and add 5ml of normal drinking water to this and rinse their mouth for 3mins with this solution and spit it out at the end. This was done morning and evening for 14 days.
  Group 1: Maintained adequate plaque control levels using mechanical methods + N.sativa oil (5ml oil + 5ml water) pulling for 3 mins twice daily in the morning and at night (after brushing/breakfast in the morning, and after brushing and before sleeping at night).
  Unified oral hygiene instructions and instructions for each intervention were provided to all participants.
  Interventions: Other: Nigella Sativa oil
- Group 2 / Chlorohexidine / CHX (Active Comparator): Group 2- Chlorohexidine (CHX).
  Chlorohexidine (Middle East Pharmaceutical Industries Ltd, Riyadh, Kingdom of Saudi Arabia).
  Each participant was given a 3 week supply of chlorohexidine. They were asked to use 10ml of CHX morning and evening, rinsing their mouth for 3 mins and then spit it out at the end. This was done morning and evening for 14 days.
  Group2: maintained adequate plaque control levels using mechanical methods + chlorohexidine rinse twice daily 10ml in the morning and at the night (after brushing/breakfast in the morning, and after brushing and before sleeping at night).
  Unified oral hygiene instructions and instructions for each intervention were provided to all participants.
  Interventions: Drug: Chlorhexidine mouthwash

INTERVENTIONS:
Other: Nigella Sativa oil — 5ml Nigella Sativa oil mixed into 5ml water prior to use and rinsed in the mouth for 3 mins and spitted out, used twice a day; morning and evening.
  Arms: Group 1 / Nigella Sativa oil / NS
Drug: Chlorhexidine mouthwash — 10ml of chlorohexidine mouthwash used for 3mins and spit out, used twice a day; morning and evening.
  Arms: Group 2 / Chlorohexidine / CHX

SUMMARY:
A double-blind randomized clinical trial was conducted for 14 days with 37 systemically healthy patients having chronic generalized gingivitis. The current study was designed to investigate the anti-inflammatory and antimicrobial efficacy of Nigella Sativa oil compared with chlorohexidine; assessing clinical parameters and gingival interleukin 6 (IL6) and interleukin 18 (IL18) levels and supra-gingival plaque analysis.

DETAILED DESCRIPTION:
A total of 37 systemically healthy patients, aged between 20 to 40 years with chronic generalised gingivitis were recruited based on the inclusion and exclusion criteria, from the Dental Clinic at Princess Nourah bint Abdulrahman University. The sample size was based on previously reported studies conducted to assess gingival crevicular interleukin levels using mouthwashes. A study information sheet was provided to each patient and the methodology of the clinical trial was explained. Written informed consent was obtained from each participant before enrolling on the study.

A double-blind randomized clinical trial was conducted Ethical clearance was obtained from the Institutional Review Board at Princess Nourah bint Abdulrahman University (Registration number: 20-0261).

Subjects were assigned computer-generated random numbers and were blindly assigned to one of two groups; Group 1- Nigella Sativa (NS) or Group 2- Chlorohexidine (CHX) (n=20) according to the sequence of the computer-generated random numbers by an investigator not directly involved in the clinical examination and sample collection. The interventions were either N. sativa oil (Al-Hussan Food Products Factory, Riyadh, Kingdom of Saudi Arabia), which was brought from the local market in Riyadh or Chlorohexidine (Middle East Pharmaceutical Industries Ltd, Riyadh, Kingdom of Saudi Arabia). Group 1: Maintained adequate plaque control levels using mechanical methods + N.sativa oil (5ml oil + 5ml water) pulling for 3 mins twice daily in the morning and at night, and Group 2: maintained adequate plaque control levels using mechanical methods + chlorohexidine rinse twice daily 10ml in the morning and at the night.

Unified oral hygiene instructions and instructions for each intervention were provided to all participants. A 24-hour contact number was provided to each participant, to report any concerns, adverse reactions or for any further information. Participants were told that they were free to drop out at any time.

Oral prophylaxis was performed on the same day of recruitment to bring the plaque score to almost zero, and the subjects in each group were given either N.sativa oil or chlorohexidine according to the blind randomised allocation by a third person. On day zero (baseline) of the trial after scaling, and on day 15 at the end of the trial; the following clinical parameters were assessed; plaque index (PI) and gingival index (GI) and plaque samples, as well as gingival crevicular fluid (GCF) samples, were collected.

Prior to the study, two dental examiners were calibrated to measure PI and GI, to reduce inter-examiner variability.

The collected data were analyzed using Graphpad PRISM (San Deigo, USA). Non-parametric signed Rank tests and parametric t-tests were used, as well as Fisher's exact test for contingency analysis. P values were calculated and a p value below 0.05 was deemed as a significant difference.

ELIGIBILITY:
Inclusion Criteria:

* At least 20 natural teeth
* Patients with moderate to severe gingivitis
* No tooth attachment loss

Exclusion Criteria:

* Periodontitis
* Cigarette smokers
* Antibiotic therapy (within the last 3 months)
* Systemic diseases
* Pregnant women
* Lactating women
* Current orthodontic treatment
* Using an intra-oral artificial prosthesis
* Using other chemical agents as a mouthwash

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Gingival index | Day 0 and day 15
Plaque index | Day 0 and day 15
IL-6 levels | Day 0 and day 15
  Measurement of IL-6 in GCF samples
IL-18 levels | Day 0 and day 15
  Measurement of IL-18 in GCF samples

SECONDARY OUTCOMES:
Bacterial load | Day 0 and day 15
  Colony forming units (CFU) count
Inhibition of types of bacterial growth | Day 0 and day 15
  Assessment on the types of bacteria present within the alpha-hemolytic class of oral bacteria

OTHER OUTCOMES:
Feedback on any adverse effects and likes/dislikes of the intervention from participants | Day 15
  Questionnaire to report on adverse effects and likes/dislikes of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ishrat Rahman, Study Director — Princess Nourah Bint Abdulrahman University
Locations (1):
- Princess Nourah bint Abdulrahman University Dental Clinic, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
At this moment in time, there is no intention or need to make individual participant data available to other researchers.